CLINICAL TRIAL: NCT02537015
Title: An Open-label Extension (OLE 2) Study to Evaluate the Safety of the 13 mg Bimatoprost Ocular Insert in Subjects With Open-angle Glaucoma or Ocular Hypertension Who Have Completed Study FSV5-004
Brief Title: An Open-label Extension Study to Evaluate the Safety of the 13 mg Bimatoprost Ocular Insert
Acronym: OLE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSV5-005 OLE 2
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Primary Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 13 mg Bimatoprost Ocular Insert (Experimental): 13 mg Bimatoprost Ocular Insert in each eye used continuously for 12 weeks, then replaced with a new 13 mg Bimatoprost Ocular Insert in each eye used continuously for another 26 weeks.
  Interventions: Drug: Bimatoprost

INTERVENTIONS:
Drug: Bimatoprost — Bimatoprost Ocular Insert in each eye used continuously for 12 weeks, then replaced with a new Bimatoprost Ocular Insert in each eye used continuously for another 26 weeks.
  Other Names: "Lumigan" is the branded name of bimatoprost in eye drop form

SUMMARY:
This study evaluated the long-term (9-months) safety of the Bimatoprost Ocular Insert in participants with Glaucoma or Ocular Hypertension who completed study FSV5-004. All the participants received Bimatoprost Ocular Insert and wore it for approximately 3 months (12 weeks), then had that Insert removed and a new Insert placed for another 26 weeks (approximately 6 months).

ELIGIBILITY:
Inclusion Criteria:

1. Completed FSV5-004 study.
2. Written informed consent prior to any study procedure.
3. Willingness to comply with the visit schedule.

Key Exclusion Criteria:

1. Participation in an investigational drug or device study other than FSV5-004 within the past 6 months or anticipated participation during the study period.
2. Subjects who will require contact lens use during the study period.
3. Any condition or situation (such as uncontrolled systemic disease) that, in the Investigator's opinion, might confound the results of the study, may put the subject at significant risk or might interfere with the subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chen, PhD, Study Director — Allergan
Locations (9):
- United States (9):
  - Vold Vision, Fayetteville, Arkansas
  - Sall Medical Research Center, Artesia, California
  - Eye Research Foundation, Newport Beach, California
  - Clayton Eye Center, Morrow, Georgia
  - Mundorf Eye Center, Charlotte, North Carolina
  - Cornerstone Health Care; Cornerstone Eye Care, High Point, North Carolina
  - University Eye Specialists, Maryville, Tennessee
  - Total Eye Care, Memphis, Tennessee
  - R&R Eye Research, LLC, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the Phase 2 study FSV5-004 [NCT02358369] were eligible to enroll in this open-label extension study.
Period: Overall Study
Arm/Group | 13 mg Bimatoprost Ocular Insert
Started | 81
Completed | 75
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Other Miscellaneous Reasons | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who had at least one Bimatoprost Ocular Insert 13 mg placed.
Arm/Group | 13 mg Bimatoprost Ocular Insert
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ocular and Non-ocular Adverse Events (AE) by Severity
Description: An AE was defined as any untoward medical occurrence (eg, sign, symptom, disease, syndrome, intercurrent illness) that occurred in a study participant, regardless of the suspected cause during the study. An ocular AE is an AE that occurred in the eye and non-ocular is an AE that occurred not in the eye. The investigator assessed the worst severity of each AE as: Mild=aware of sign or symptom, but readily tolerated, Moderate=discomfort enough to cause interference with usual activity or Severe=incapacitating with inability to work or do usual activity.
Time Frame: Baseline (Day 0, enrollment in this study) to end of study (Week 38)
Population: Safety Population included all enrolled participants who had at least one 13 mg Bimatoprost Ocular Insert placed.
Measure: Number; unit: percentage of participants
Arm/Group | 13 mg Bimatoprost Ocular Insert
Number analyzed (Participants) | 81
percentage of participants
  Ocular, Mild | 25.9
  Ocular, Moderate | 11.1
  Ocular, Severe | 0
  Non-Ocular, Mild | 6.2
  Non-Ocular, Moderate | 8.6
  Non-Ocular, Severe | 4.9

2. Other Pre Specified Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. IOP measurements were taken at 8 am (Time (T)=0 hour) at Weeks 4, 8, 12, 24 and 38. Diurnal IOP measurements were also taken at 10 am (T=2 hour), and 4 pm (T=8 hour) at Weeks 12, 24 and 38. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated an improvement. Baseline is defined as the IOP assessment done at the Randomization visit (Day 0) of study FSV5-004.
Time Frame: Baseline (Day 0 in study FSV5-004) to Weeks 4, 8, 12, 24 and 38
Population: Per Protocol, this Outcome Measure previously registered on ClinicalTrials.gov as a Secondary Outcome Measure is an Other Pre-specified Outcome Measure.
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Percentage of Participants by Subject-Reported Comfort Assessment Categories
Description: The participant assessed their overall comfort with ocular inserts using the following rating choices: Not aware of inserts, very comfortable; Aware of inserts, and comfortable; Tolerable, but mild discomfort; Moderate discomfort or Severe discomfort. The percentage of participants in each rating category is reported.
Time Frame: Baseline (Day 0, enrollment in this study) Weeks 4, 8, 12, 24 and 38
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Bimatoprost Ocular Insert Retention Duration
Description: Insert duration was defined as the total duration (in days) that any ocular insert remained in place for each subject, measured from the date of Insert removal minus date of Insert placement + 1.
Time Frame: Baseline (Day 0, enrollment in this study) to the end of study (Week 38)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Percentage of Participants Who Received Rescue Treatment
Description: Rescue treatment with topical bimatoprost was available for each eye if deemed necessary by the investigator to achieve desired IOP.
Time Frame: Baseline (Day 0, enrollment in this study) to the end of study (Week 38)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change From Baseline in Endothelial Cell Count
Description: Density (number of cells/mm^2) of corneal endothelial cells was determined at four sites using specular microscopy of the central corneal endothelium at Baseline and at Week 38.
Time Frame: Baseline (Day 0, enrollment in this study) to end of study (Week 38)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline (Day 0-enrollment in this study) to the end of study (Week 38)
Arm/Group | 13 mg Bimatoprost Ocular Insert
Serious Adverse Events (participants affected / at risk) | 7/81
Other Adverse Events (participants affected / at risk) | 20/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13 mg Bimatoprost Ocular Insert (N=81)
Atrial fibrillation (Cardiac disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 13 mg Bimatoprost Ocular Insert (N=81)
Punctate keratitis (Eye disorders) | 10
Eye discharge (Eye disorders) | 9
Ocular discomfort (Eye disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No presentation or publication of Institution's data relating to the Trial may occur until after the Trial has been completed at all sites. If Investigator desires to present or publish, investigator must submit any and all manuscripts, posters, abstracts, or other intended publications (hereinafter collectively referred to as "manuscripts") to Sponsor at least sixty (60) days prior to the actual submission of such manuscript(s) for publication.